CLINICAL TRIAL: NCT04146545
Title: CommunityRx-Dementia: A Study for Primary Caregivers of Loved Ones With Alzheimer's Disease and Related Dementias
Brief Title: CommunityRx-Dementia
Acronym: CRx-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB20-0301; 1R01AG064949-01 (NIH)
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Health Related Social Needs (HRSN)
Keywords: caregivers; dementia; information-sharing; Alzheimer's Disease; caregiving; community resources
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Cases will receive the CRx-D Intervention. Controls will not receive the intervention but will receive the usual standard of care.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Experimental): Community Rx-Dementia "CRxD" Caregiver Resources
  Interventions: Behavioral: Community Rx-Dementia "CRxD" Caregiver Resources
- Control (No Intervention): Usual Standard Care

INTERVENTIONS:
Behavioral: Community Rx-Dementia "CRxD" Caregiver Resources — A tailored list of resources addressing health-related social needs (HRSN) for caregivers and access to an online community resource finder.
  Other Names: CRx-D
  Arms: Cases

SUMMARY:
Caregivers of home-dwelling people with Alzheimer's Disease and related dementias (ADRD) are one of the most rapidly growing populations in the United States. Among ADRD caregivers with unmet health-related social needs, this study aims to evaluate the effects of the CRx-D intervention versus usual care on caregiver self-efficacy.

DETAILED DESCRIPTION:
The CRx-D intervention is a caregiver-centered adaptation of CommunityRx (CRx), an information-based intervention that systematically matches people to nearby community resources for health-related social needs. We are conducting a single-blind randomized controlled trial and enrolling caregivers through UChicago-affiliated clinic sites. Caregivers will be screened and asked about unmet health-related social needs at the outpatient visit. Eligible, self-identified caregivers will complete an in-person baseline survey on-site (face to face), followed by phone surveys at 7, 30, 90 days, and 12 months. Caregivers randomized to the intervention will receive tailored information on community resources for their identified health-related social needs. They will also be given access to an online community-resource tool and shown how to use it, so they can search for additional resources in their community beyond the point-of-care and outside of the clinic. All caregivers (regardless of research arm) will also receive a series of text messages related to the study such as reminders to schedule the phone survey with a member of the research team.

The anticipated sample (n=414) includes pretest participants (n=20), RCT participants enrolled in the 12-month RCT (n=344) and additional men caregivers enrolled in a 3-month RCT (N=50).

ELIGIBILITY:
Inclusion Criteria:

* Resides in the target geographic region of the study (living in 1 of the 35 target zip codes)
* Self-identifies as a caregiver of a home-dwelling person with Alzheimer's Disease or related dementia using an adaptation of the BRFSS caregiver module
* Has access to a cell phone and provides the research interviewer with the cell phone number
* Agrees to receive text messages from the study
* Has a personal email address.
* Self-report their gender identity to be male or trans male/trans man (only for additional 50 caregivers enrolled in the 3-month RCT)

Exclusion Criteria:

* Past enrollment in the CommunityRx-C study
* Recollection of previous receipt of a HealtheRx

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Abramsohn EM, De Ornelas M, Borson S, Frazier CRM, Fuller CM, Grana M, Huang ES, Jagai JS, Makelarski JA, Miller D, Schulman-Green D, Shiu E, Thompson K, Winslow V, Wroblewski K, Lindau ST. CommunityRx, a social care assistance intervention for family and friend caregivers delivered at the point of care: two concurrent blinded randomized controlled trials. Trials. 2023 Oct 21;24(1):681. doi: 10.1186/s13063-023-07697-z. PMID 37864258
- [Derived] Abramsohn EM, De Ornelas M, Borson S, Frazier CR, Fuller CM, Grana M, Huang ES, Jagai JS, Makelarski JA, Miller D, Schulman-Green D, Shiu E, Thompson K, Winslow V, Wroblewski K, Lindau ST. Two concurrent randomized controlled trials of CommunityRx, a social care intervention for family and friend caregivers delivered at the point of care. Res Sq [Preprint]. 2023 Mar 1:rs.3.rs-2464681. doi: 10.21203/rs.3.rs-2464681/v1. PMID 36909590

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cases | Control
Started | 178 | 182
Main Randomized Trial (These were the participants enrolled in the main randomized trial as proposed in the original grant.) | 171 | 173
Supplement (Additional supplemental funding was obtained to enrich the sample with male caregivers and 16 additional participants were enrolled and followed for 3 months) | 7 | 9
Completed | 177 | 182
Not Completed | 1 | 0
Not completed — deemed ineligible after randomization | 1 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants except for 1 who was deemed ineligible after randomization
Groups:
- Cases - Main Randomized Trial: Community Rx-Dementia "CRxD" Caregiver Resources, Enrolled as part of the Main Randomized Trial
  Community Rx-Dementia "CRxD" Caregiver Resources: A tailored list of resources addressing health-related social needs (HRSN) for caregivers and access to an online community resource finder.
- Control - Main Randomized Trial: Usual Standard Care - Enrolled as part of the Main Randomized Trial
- Cases - Supplement: Community Rx-Dementia "CRxD" Caregiver Resources, Enrolled as part of the Supplement
  Community Rx-Dementia "CRxD" Caregiver Resources: A tailored list of resources addressing health-related social needs (HRSN) for caregivers and access to an online community resource finder.
- Control - Supplement: Usual Standard Care - Enrolled as part of the Supplement
- Total: Total of all reporting groups
Arm/Group | Cases - Main Randomized Trial | Control - Main Randomized Trial | Cases - Supplement | Control - Supplement | Total
Number analyzed (Participants) | 170 | 173 | 7 | 9 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.8) | 59.0 (12.0) | 58.7 (15.3) | 58.6 (13.5) | 59.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed differs from overall due to missing data
  Participants
    number analyzed (Participants) | 169 | 173 | 7 | 9 | 358
    Female | 133 | 135 | 0 | 0 | 268
    Male | 36 | 38 | 7 | 9 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Number analyzed differs from overall due to missing data
  Participants
    Non-Hispanic Black: number analyzed (Participants) | 170 | 170 | 7 | 9 | 356
    Non-Hispanic Black | 142 | 132 | 7 | 5 | 286
    Non-Hispanic White: number analyzed (Participants) | 170 | 170 | 7 | 9 | 356
    Non-Hispanic White | 11 | 16 | 0 | 3 | 30
    Hispanic: number analyzed (Participants) | 170 | 170 | 7 | 9 | 356
    Hispanic | 7 | 7 | 0 | 1 | 15
    Other: number analyzed (Participants) | 170 | 170 | 7 | 9 | 356
    Other | 10 | 15 | 0 | 0 | 25
Region of Enrollment [Number; unit: participants]
  United States | 170 | 173 | 7 | 9 | 359
Presence of at least 1 health-related social risk factor [Count of Participants; unit: Participants] — Presence of at least one health-related social risk factor (HRSR) at baseline based on the Accountable Health Communities screening tool, including food, housing, transportation, utilities, and safety. Standard scoring guidelines were used and participants' baseline HRSR status was categorized as none versus one or more HRSRs.
  Participants
    None | 106 | 104 | 5 | 4 | 219
    One or more | 64 | 69 | 2 | 5 | 140

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Self-efficacy at 12 Months Among Caregivers With Unmet Health Related Social Needs
Description: Self-efficacy is measured with a 4-item sub-domain from the 2015 Caregiver Dementia Care and Self-Efficacy Survey (Jennings et al). Responses to each of the items are scored between 1 = "strongly disagree" to 5 = "strongly agree" and will generate an average score. Higher values = greater self-efficacy
Time Frame: 12 months
Population: Analysis was restricted to caregivers in the main randomized trial who had at least 1 unmet health-related social need at baseline and completed the self-efficacy measure at 12 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cases | Control
Number analyzed (Participants) | 39 | 36
score on a scale | 3.5 (0.7) | 3.5 (1.0)

2. Primary Outcome: Satisfaction With Care
Description: Satisfaction will be assessed using the Patient Satisfaction Questionnaire 18-item short form (PSQ-18), specifically the general satisfaction sub-scale (2 questions). Five possible response options for each of the two items are scored 1 to 5; with a higher score equating to higher satisfaction. Scores will be transformed using the formula: y= 100 * (x-a)/(b-a) where y=the transformed score, x=the original score, a=the minimum possible score and b=the maximum possible score. Transformed items will be averaged to generate the composite score (range 0-100; higher scores indicating greater satisfaction).
Time Frame: 7 days
Population: Analysis was restricted to caregivers in the main randomized trial who completed the satisfaction measure at 1 week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cases | Control
Number analyzed (Participants) | 160 | 156
score on a scale | 71.4 (19.3) | 69.6 (21.8)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Cases | Control
All-Cause Mortality (participants affected / at risk) | 0/177 | 0/182
Serious Adverse Events (participants affected / at risk) | 0/177 | 0/182
Other Adverse Events (participants affected / at risk) | 0/177 | 0/182

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT04146545/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT04146545/SAP_001.pdf
  • Informed Consent Form (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT04146545/ICF_002.pdf